CLINICAL TRIAL: NCT03993249
Title: Nivolumab Plus Chemoradiotherapy in Patients With Muscle-invasive Bladder Cancer (MIBC) Not Undergoing Cystectomy: a Phase II, Randomized Study
Brief Title: Nivolumab Plus Chemoradiotherapy in Patients With Muscle-invasive Bladder Cancer (MIBC) Not Undergoing Cystectomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hellenic GenitoUrinary Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REQ-0000020479
Record Dates: First submitted 2019-06-04; First posted 2019-06-20 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Nivolumab; Chemoradiotherapy

STUDY DESIGN:
Intervention Model Description: randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemoradiotherapy (Other): standard of care chemo-radiotherapy
  Interventions: Other: chemoradiotherapy
- Combination (Experimental): standard of care chemo-radiotherapy + Nivolumab
  Interventions: Biological: Nivolumab; Other: chemoradiotherapy

INTERVENTIONS:
Biological: Nivolumab — standard of care chemoradiotherapy + Nivolumab
  Arms: Combination
Other: chemoradiotherapy — standard of care chemoradiotherapy

SUMMARY:
The purpose of this study is to investigate the effect synchronous use of nivolumab in addition to chemoradiotherapy in patients withnon-metastatic MIBC who are not candidates for radical cystectomy

DETAILED DESCRIPTION:
The initial hypothesis is that addition of nivolumab will increase 2-year locoregional control rate from 55% (control arm) to 75% (immunotherapy arm)

There is a 24 month accrual period during which 78 patients will be randomized in a control group (standard chemo-radiotherapy) and the treatment group (chemo-radiotherapy + Nivolumab)

The primary objective would be to compare locoregional control rate at 2-years between patients with MIBC receiving or not receiving nivolumab in addition to chemoradiotherapy.

The secondary objectives are

1. To study the safety of the addition of nivolumab to chemoradiotherapy in patients with MIBC
2. To compare 2-year bladder cancer failure-free (BCFF) rates, defined as distant metastasis free survival (MFS) AND/OR locoregional failure (defined as in primary objective)
3. To compare median overall survival (OS) in patients with MIBC receiving or not receiving nivolumab in addition to chemoradiotherapy
4. Assess the effect of combined treatment on the quality of life

Correlative studies of outcomes with PD-L1expression and with lymphocytic populations in the environment of the tumor

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, muscle-invasive carcinoma of the bladder, cT2-T4aN0M0
* Urothelial, squamous or glandular histology according to WHO 2016 classification (Fig 1)
* Undergone a vigorous TURB
* Not candidates for radical cystectomy.
* PS:0-1
* age >18 years old
* Adequate bone marrow function
* Adequate renal function

Exclusion Criteria:

Key Exclusion Criteria

* Histology other than transitional-cell, squamous or adenocarcinoma
* Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, prostate cancer cervix or breast.
* Previous systemic chemotherapy or prior biologic agents within 4 weeks, or intravesical Bacillus Calmette-Guerin (BCG) within 6 weeks of the first dose of study treatment.
* Prior treatment with any PD-1 or PDL-1 inhibitor or anti CTLA4 agent
* Previous pelvic radiation therapy.
* Patients with inherited syndromes associated with hypersensitivity to ionizing radiation
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation
* Any history of inflammatory bowel disease and or history of abdominal fistula
* Previous allergy to any of the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-05-28 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Locoregional control rate | 2 years
  To compare locoregional control rate at 2-years between patients with MIBC receiving or not receiving nivolumab in addition to chemoradiotherapy

SECONDARY OUTCOMES:
Incidence Rate of treatment-related adverse event (safety and tolerability) | 2 years
  Incidence of adverse events as assessed by CTCAE. After radiotherapy completion, AEs will be assessed according to RTOG/EORTC Late Radiation Morbidity Scoring Schema
Bladder cancer failure-free (BCFF) rates | 2 years
  To compare 2-year bladder cancer failure-free (BCFF) rates, defined as distant metastasis free survival (MFS) AND/OR locoregional failure (defined as in primary objective)
Median overall survival (OS) | 2 years
  To compare median overall survival (OS) in patients with MIBC receiving or not receiving nivolumab in addition to chemoradiotherapy
Assessment of the effect of the combined treatment on the quality of life | 2 years
  Quality of life score assessed by Quality of Life of Cancer Patients Questionnaire (EORTC QLQ-C30). Discomfort measured in a scale from 1 (not at all) to 4 (very much) Overall health and quality of life score measured in a scale from 1 (very poor) to 7 (excellent)

CONTACTS AND LOCATIONS:
Locations (1):
- Hellenic GenitoUrinary Cancer Group, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No